CLINICAL TRIAL: NCT06002438
Title: Egg to Ameliorate Environmental Enteric Dysfunction and Improve Growth in Children With Moderate Acute Malnutrition
Brief Title: Eggs for Gut Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Project Peanut Butter (Other); Thrasher Research Fund (Other); Ministry of Health and Sanitation, Sierra Leone (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202306090
Record Dates: First submitted 2023-08-10; First posted 2023-08-21 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Moderate Acute Malnutrition; Stunting; Environmental Enteric Dysfunction; Severe Acute Malnutrition
MeSH Terms: conditions — Growth Disorders; Severe Acute Malnutrition | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The intervention and control powders will be packaged such that investigators and outcomes assessors will not know their identity. Participants and care providers are likely to be able to distinguish them, however.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg powder (Experimental): 15g egg powder per day for 24 weeks
  Interventions: Dietary Supplement: Whole egg powder; Dietary Supplement: Supercereal Plus; Dietary Supplement: Micronutrient sprinkles; Drug: Sulfadoxine pyrimethamine
- Corn powder (Active Comparator): 15g corn powder per day for 24 weeks
  Interventions: Dietary Supplement: Corn powder; Dietary Supplement: Supercereal Plus; Dietary Supplement: Micronutrient sprinkles; Drug: Sulfadoxine pyrimethamine

INTERVENTIONS:
Dietary Supplement: Whole egg powder — 15g daily dose for 24 weeks
  Arms: Egg powder
Dietary Supplement: Corn powder — 15g daily dose for 24 weeks
  Arms: Corn powder
Dietary Supplement: Supercereal Plus — Approximately 110 g per day (1.5 kg every 2 weeks) supplementary food to be provided for treatment of MAM for up to 6 weeks.
Dietary Supplement: Micronutrient sprinkles — To be provided after completion of MAM supplementary feeding. Provides 1 RDA of 14 micronutrients.
Drug: Sulfadoxine pyrimethamine — Infants < 12 months of age: 250/12.5mg SP at enrollment, week 6, week 12, week 18.
  Infants >= 12 months of age: 500/25mg SP at enrollment, week 6, week 12, week 18.
  Other Names: SP

SUMMARY:
The goal of this clinical trial is to test egg powder supplementation in children with moderate acute malnutrition in Sierra Leone. The main question it aims to answer is:

- Will provision of 15g of whole egg powder per day during and after treatment for moderate acute malnutrition (for 24 weeks total) improve small intestinal permeability and linear growth among 6-30 month old Sierra Leonean children compared with daily corn powder supplementation?

DETAILED DESCRIPTION:
Undernutrition in children manifests as wasting, stunting, or both. While wasting is generally responsive to high-quality nutritional interventions, stunting is less so. Affected children are at increased risk of acute and chronic illnesses, have reduced neurocognitive development, lower academic achievement, reduced adult earning potential, and shortened lifespans. Given that stunting affects over 140 million children at any one time, the costs incurred are deep and broad, particularly among children in sub-Saharan Africa, where nearly half of the world's population growth is expected to occur over the next 30 years. Part of the challenge of treating stunting has been attributed to environmental enteric dysfunction (EED), an acquired small intestine disorder characterized by chronic inflammation, villus blunting, and impaired nutrient absorption. EED is prevalent in the same populations plagued by stunting, develops concurrently with loss in linear growth, and has explained upwards of 43% of observed growth faltering. EED has recently also been found in over 75% of children with moderate acute malnutrition (MAM, moderate wasting) in Sierra Leone, a population with high rates of deterioration to severe acute malnutrition and death, 20%. EED is a plausible cause for this treatment resistance, and for the high rates of recurrence seen in these children. There is an urgent need to increase understanding of the concurrence of stunting, EED, and wasting, and to test interventions targeted to their pathological underpinnings. Dietary egg can play a critical role in the fight against malnutrition by providing abundant high-quality protein and nutrients essential for physical and cognitive recovery. One egg/day has been shown to reduce stunting in several contexts. Recent evidence has shown that short-term egg/bovine colostrum supplement given to 9-12-month-old Malawian children improved linear growth and intestinal permeability in children with severe EED. It is possible that prolonged supplementation with egg in a high-risk population in rural Sierra Leone could improve acute and long-term health trajectories for children and put eggs on the map for food aid. This will be a randomized, investigator-blinded, controlled clinical trial testing whether daily supplementation with 15g whole egg powder during and for 18 weeks after treatment for moderate acute malnutrition might reduce intestinal permeability and improve linear growth, among other outcomes, when compared with control corn powder. Children with relatively higher risk MAM will be enrolled (MUAC < 12.5 cm AND MUACz < -2), treated with Supercereal Plus for up to 6 weeks, and undergo urine and stool collections at 6, 12, and 24 weeks. Urine collections will be for assessment of lactulose permeability and will involve participant consumption of a known amount of lactulose and collection of all urine over at least 4 hours thereafter. Stool collections will be for fecal host mRNA transcripts and selected proteins. Participants will also receive intermittent malaria chemoprophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months of age and less than 30 months of age
* Mid-upper arm circumference >= 11.5cm and < 12. 5 cm
* Mid-upper arm circumference-for-age z-score < -2
* Provision of signed (or thumb-printed) and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study, including no plan to move from the catchment area of a participating clinic

Exclusion Criteria:

* Nutritional edema
* Simultaneous involvement in another research trial or supplementary feeding program
* Chronic debilitating illness
* Allergy to egg
* Receipt of treatment for acute malnutrition within 1 month prior to screening

Ages: 6 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 461 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Percent lactulose excretion | Collected 12 and 24 weeks after enrollment
  Percent lactulose excretion in urine over >=4 hours after lactulose consumption
Change in length-for-age z-score | To be compared at 12 and 24 weeks after enrollment
  Difference in length-for-age z-score between enrollment and weeks 12 and 24

SECONDARY OUTCOMES:
Percent Lactulose excretion >= 0.2 and >=0.45 | Collected 6, 12, and 24 weeks after enrollment
  Proportion with moderately and severely abnormal small intestinal permeability. Percent lactulose excretion in urine over >=4 hours after lactulose consumption
Rate of length gain | Across 24 week follow-up period
  mm/week
LAZ < -2 | To be compared at 12, 18, and 24 weeks after enrollment
  Proportion stunted
Fecal host mRNA transcripts | Collected 12 and 24 weeks after enrollment
  CD53, CDX1, HLA-DRA, TNF, S100A8, MUC12, and REG1A
Fecal host protein alpha-1 antitrypsin | Collected 12 and 24 weeks after enrollment
  Level of alpha-1 antitrypsin, mg/g
Fecal host protein myeloperoxidase | Collected 12 and 24 weeks after enrollment
  Level of myeloperoxidase, ng/mL
Fecal host protein neopterin | Collected 12 and 24 weeks after enrollment
  Level of neopterin, nmol/L
Rate of weight gain | Enrollment to week 6 (MAM treatment phase), and across 24 week follow-up period
  g/kg/d
Percent Lactulose excretion | 6 weeks after enrollment
  Percent lactulose excretion in urine over >=4 hours after lactulose consumption
Deterioration to severe acute malnutrition | Time-to-event across follow-up period
  Mid-upper arm circumference < 11.5 cm and/or nutritional edema
Recurrence of MAM | Time-to-event across follow-up period
  Development of MUAC < 12.5 cm among those who achieved MUAC >= 12.5 cm during initial MAM treatment
Sustained recovery | Across 24 week follow-up period
  Defined by achievement mid-upper arm circumference >= 12.5 cm without nutritional edema and maintenance of MUAC >= 12.5 cm throughout follow-up thereafter.
Death | Time-to-event across follow-up period
  As defined by caregiver report
Graduation | Within 6 weeks of enrollment
  Defined by mid-upper arm circumference >= 12.5 cm

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (10):
- Sierra Leone (10):
  - Bandajuma, Bandajuma, Southern Province
  - Bendu Maleh, Bendu, Southern Province
  - Blama Massaquoi, Blama Massaquoi, Southern Province
  - Gbondapi, Gbondapi, Southern Province
  - Gofor, Gofor, Southern Province
  - Jendema, Jendema, Southern Province
  - Potoru, Potoru, Southern Province
  - Pujehun Static, Pujehun, Southern Province
  - Taninahun, Taninahun, Southern Province
  - Zimmi, Zimmi, Southern Province

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of primary publication

REFERENCES:
- [Derived] Stephenson KB, Greenfeld A, Ryan MG, Kleban E, Kwak L, Lee A, Wegner DR, Jiang X, Hendrixson DT, Kamara MT, Koroma AS, Manary MJ. Egg supplementation for 24 weeks does not improve linear growth or reduce small intestinal permeability in Sierra Leonean children with moderate wasting: a randomized, blinded, controlled trial. Am J Clin Nutr. 2025 Nov;122(5):1326-1337. doi: 10.1016/j.ajcnut.2025.08.019. Epub 2025 Oct 14. PMID 41193034